CLINICAL TRIAL: NCT06058455
Title: A Randomized Controlled Trial of the Efficacy of IDEA3 - An Evidence-based Sexual Assault Resistance Intervention for Undergraduate Women Adapted for Internet Delivery
Brief Title: An Evaluation of an Online Sexual Assault Resistance Program (IDEA3)
Acronym: IDEA3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: University of Windsor (Other); University of Nebraska (Other); University of Guelph (Other); Tufts University (Other); University of Central Florida (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Sarah Peitzmeier, Associate Professor of Behavioral and Community Health, University of Maryland, College Park
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00229565; 23-063 (Other: UWindsor REB (responsible REB)); 183649 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2023-09-12; First posted 2023-09-28 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Sexual Assault

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IDEA3 sexual assault resistance intervention (Experimental): IDEA3 curriculum will be delivered by pairs of trained facilitators over Zoom to reach up to 8 pairs of female-identified university students in four, 3-hour units. The four units will be spread over two to four weeks' time.
  Interventions: Behavioral: IDEA3 Sexual Assault Resistance Intervention
- Consent workshop (Active Comparator): Randomized participants who do not receive the intervention will receive one 60-minute session consisting of an internet delivered (Zoom) consent workshop.
  Interventions: Behavioral: Consent Workshop

INTERVENTIONS:
Behavioral: IDEA3 Sexual Assault Resistance Intervention — Internet-delivered EAAA (IDEA3), adapted from an in-person sexual assault resistance education intervention: Enhanced Assess, Acknowledge, Act (EAAA) intervention that was found in a randomized trial to reduce sexual assault victimization by about 50% at follow-up. IDEA3 designed for female identifying university students and focuses on resisting sexual assault committed by males in 4, 3-hour units: 1-ASSESS builds ability to detect risk with male acquaintances and develop risk reduction strategies. 2-ACKNOWLEDGE explores overcoming emotional barriers preventing women from acknowledging risk and employing effective resistance strategies with males. 3-ACT shows effectiveness of resistance strategies and teaches verbal and physical self-defense in common situations. 4-RELATIONSHIPS & SEXUALITY adapts the Our Whole Lives curriculum to increase women's comfort in talking about sex/sexuality and identify sexual values/desires.
  Arms: IDEA3 sexual assault resistance intervention
Behavioral: Consent Workshop — Participant pairs assigned to the control arm will receive a 60-minute session consisting of a 60-min interactive, virtual consent workshop. The workshop will include information on a) what consent is, including the idea that consent is about bodily autonomy and applies to interactions beyond sex, b) how to give and ask for consent, and c) examples of what it looks like to ask for and give/not give consent. This presentation will be given by a well-trained Research Assistant.
  Arms: Consent workshop

SUMMARY:
The goal of this randomized trial is to test whether the Internet-Delivered Enhanced Assess, Acknowledge, Act (IDEA3) sexual assault resistance education intervention reduces sexual violence victimization in undergraduate women.

Participants in the intervention group will be asked to attend four three-hour group sessions of a sexual assault resistance program called IDEA3 with a partner, as well as fill out a number of surveys. Participants in the control group will be asked to attend a one-hour consent workshop with a partner and fill out surveys.

Researchers will compare sexual assault victimization between the groups in the one year following the intervention.

DETAILED DESCRIPTION:
Sexual violence (SV), which occurs along a continuum from unwanted sexual contact to rape, is common among young women, with some 40% experiencing sexual assault during their time in college. Given the numerous negative consequences associated with SV, developing effective SV prevention and resistance programs for young adult women is critical for reducing victimization and improving health outcomes for adolescent girls. The Enhanced Assess, Acknowledge, Act (EAAA) sexual assault resistance program has been shown to substantially reduce rates of SV (50% for rape and attempted rape) in young women attending university (ages 17-24). The purpose of the current study is to test the efficacy of the newly adapted Internet-Delivered Enhanced Assess, Acknowledge, Act (IDEA3) program in reducing sexual violence victimization among undergraduate women over 12 months of follow-up. IDEA3 is a 12-hour psychoeducational intervention that provides information, skills, and practice aimed at a) decreasing the time needed for young women to assess sexually coercive situations as dangerous and to take action, b) reducing emotional obstacles to taking action, c) increasing the use of the most effective methods of verbal and physical self-defense, and d) identifying sexual and relationship values and boundaries and reinforcing the right to defend them.

ELIGIBILITY:
Inclusion Criteria:

* 1st- and 2nd-year university students at one of the 4 sites
* female-identifying students
* students between ages of 17-24
* able to attend one of the scheduled program groups
* able and willing to be matched with another eligible student

Exclusion Criteria:

- None

Ages: 17 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Cisgender or transgender women
Enrollment: 1920 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Completed rape | Baseline, 1-week post-intervention, 6-months and 12-months after randomization
  The Sexual Experiences Survey Short Form Victimization (SES-SFV) will be used to measure the primary sexual assault outcomes. Completed rape will have occurred when a participant indicates she has had at least one experience of threatened, forced, or drugged completed (not attempted) sexual activity (oral, anal, or vaginal intercourse - answered 'once' or more to any of 9 questions (2c, 2d, 2e, 3c, 3d, 3e, 4c, 4d, or 4e) in the period between the baseline measurement and the 12-month survey measurement.

SECONDARY OUTCOMES:
Attempted rape | Baseline, 1-week post-intervention, 6-months and 12-months after randomization
  The SES-SFV will also be used to measure secondary sexual assault outcomes: Attempted rape will have occurred when a participant indicates she has had at least one experience of threatened, forced, or drugged attempted (not completed) sexual activity (oral, anal, or vaginal intercourse - answered 'once' or more to any of 9 questions (5c, 5d, 5e, 6c, 6d, 6e, 7c, 7d, or 7e) in the period between the baseline and the 12-month survey.
Other Forms of Sexual Assault | Baseline, 1-week post-intervention, 6-months and 12-months after randomization
  The SES-SFV will also be used to measure other sexual assault outcomes:
  Non-penetrative forced sexual contact will have occurred when a participant indicates she has had at least one such experience of non-penetrative sexual contact by any perpetrator strategy - answered 'once' or more to any of 5 questions (1a, 1b, 1c, 1d, 1e).
  Completed sexual coercion will have occurred when a participant indicates she has had at least one experience of coerced (not forced) completed sexual activity (oral, anal, or vaginal intercourse - answered 'once' or more to any of 6 questions (2a, 2b, 3a, 3b, 4a, 4b).
  Attempted sexual coercion will have occurred when a participant indicates she has had at least one experience of coerced (not forced) attempted (not completed) sexual activity (oral, anal, or vaginal intercourse - answered 'once' or more to any of 6 questions (5a, 5b, 6a, 6b, 7a, 7b).

OTHER OUTCOMES:
Self-defense self-efficacy | Baseline, 1-week post-intervention, 6-months and 12-months after randomization
  Measured with a questionnaire to assess changes from baseline in women's confidence that they could defend themselves if confronted with a sexual assault situation.
Perception of personal risk | Baseline, 1-week post-intervention, 6-months and 12-months after randomization
  A single item will be used to measure women's perception of their personal risk of sexual assault by male acquaintances.
Detection of risk cues | 1-week post-intervention, 6-months and 12-months after randomization
  Participants' ability to detect risk in hypothetical assault scenarios will be assessed at the first time point by a measure in which participants read a scenario and then complete a subscale assessing their perception of the situation. At the other time points a measure will be used in which an acquaintance (6-mos) and stranger (12-mos) vignette unfolds line by line and the point at which participants indicate they would become uncomfortable and when they would leave the scenario are recorded. Receiving the same scenario/vignette more than once invalidates the measures.
Willingness to use Effective Self-Defense Strategies | 1-week post-intervention
  Using the same vignettes participants read to assess the Detection of Risk Cues outcome, the Direct Resistance scale of an untitled measure developed by Testa et al (2006) will be used to assess participants' willingness to use effective self-defense strategies at different points while reading a vignette of a sexual assault scenario.
Rape Myth Acceptance | Baseline, 1-week post-intervention, 6-months and 12-months after randomization
  The Updated Illinois Rape Myth Acceptance scale will be used to assess respondents' belief in prejudicial and false ideas about rape.
Belief in Female Precipitation of Rape | Baseline, 1-week post-intervention, 6-months and 12-months after randomization
  The female precipitation subscale of the Perceived Causes of Rape scale will be used to measure beliefs that women cause rape.
Knowledge of and Willingness to Use Effective Self-Defense Strategies | 1-week post-intervention, 6-months and 12-months after randomization
  An open-ended question will be used to measure participants' knowledge of and willingness to use of the most effective self-defense strategies at follow-ups. Participants will respond to the question "If a man I knew (e.g., a date or acquaintance) tried to force me to have sex with him when I didn't want to, I would ..." Using a coding system, these responses will be scored by two independent coders (blinded to the randomization group) for the presence or absence of effective forceful physical resistance and forceful verbal resistance strategies and their frequencies (e.g., punch, kick, and bite are all examples of forceful physical resistance).
Acceptance of Sexualized Aggression | Baseline, 1-week post-intervention, 6-months and 12-months after randomization
  Increases or decreases in acceptance of sexualized aggression will be assessed as measured by the 15-item Acceptance of Sexualized Aggression scale.
Sexual and Reproductive Empowerment Scale | Baseline, 1-week post-intervention, 6-months and 12-months after randomization
  The Sexual and Reproductive Empowerment Scale assesses sexual and reproductive empowerment among adolescents and young adults. Investigators will use 13 items from the four subscales of sexual safety; self-love; sense of future; and sexual pleasure.
Self-Blame Following Sexual Assault | Baseline, 1-week post-intervention, 6-months and 12-months after randomization
  Behavioral self-blame subscale from the Rape Attribution Questionnaire will be used to assess the extent to which women who are sexually assaulted in the follow-up timeframe of the trial blame themselves for the incident(s).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M Peitzmeier, PhD, Principal Investigator — University of Maryland; Charlene Y Senn, PhD, Principal Investigator — University of Windsor
Locations (6):
- United States (4):
  - University of Central Florida, Orlando, Florida
  - University of Maryland, College Park, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - University of Nebraska - Lincoln, Lincoln, Nebraska
- Canada (2):
  - University of Guelph, Guelph, Ontario
  - University of Windsor, Windsor, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Qualified academic researchers will be allowed to access de-identified survey responses upon request to the PIs, or a designee such as a secure data repository, e.g. ICPSR. The final system for managing and approving requests has yet to be determined.
Supporting Information: Study Protocol, SAP
Time Frame: From first publication and available for at least 5 years
Access Criteria: The final system for managing and approving requests has yet to be determined.

REFERENCES:
- [Background] Cowan, G., & Campbell, R. R. (1995). Rape causal attitudes among adolescents. Journal of Sex Research, 32(2), 145-153.
- [Background] Cowan, G., & Quinton, W. J. (1997). Cognitive style and attitudinal correlates of the perceived causes of rape scale. Psychology of Women Quarterly, 21(2), 227-245.
- [Background] Frazier PA. Perceived control and distress following sexual assault: a longitudinal test of a new model. J Pers Soc Psychol. 2003 Jun;84(6):1257-69. doi: 10.1037/0022-3514.84.6.1257. PMID 12793588
- [Background] Gray, M. D., Lesser, D., Quinn, E., & Brounds, C. (1990). The effectiveness of personalizing acquaintance rape prevention: Programs on perception of vulnerability and on reducing risktaking behavior. Journal of College Student Development, 31, 217-220.
- [Background] Marx BP, Calhoun KS, Wilson AE, Meyerson LA. Sexual revictimization prevention: an outcome evaluation. J Consult Clin Psychol. 2001 Feb;69(1):25-32. doi: 10.1037//0022-006x.69.1.25. PMID 11302273
- [Background] Messman-Moore, T. L., & Brown, A. L. (2006). Risk perception, rape and sexual revictimization: A prospective study of college women. Psychology of Women Quarterly, 30, 159-172. doi:10. 1111/j.1471-6402.2006.00279.x
- [Background] Payne, D. L., Lonsway, K. A., & Fitzgerald, L. F. (1999). Rape myth acceptance: Exploration of its structure and its measurement using the Illinois Rape Myth Acceptance Scale. Journal of Research in Personality, 33, 27-68.
- [Background] Senn, C. Y., Gee, S. S., & Thake, J. (2011). Emancipatory sexuality education and sexual assault resistance: Does the former enhance the latter?. Psychology of Women Quarterly, 35(1), 72-91.
- [Background] Papp, L. J. (2023). Sexualized aggression in college drinking settings: A four-year prospective cohort study of undergraduate women [Unpublished doctoral dissertation]. University of Michigan.
- [Background] Testa M, Vanzile-Tamsen C, Livingston JA, Buddie AM. The role of women's alcohol consumption in managing sexual intimacy and sexual safety motives. J Stud Alcohol. 2006 Sep;67(5):665-74. doi: 10.15288/jsa.2006.67.665. PMID 16847534
- [Background] Upadhyay UD, Danza PY, Neilands TB, Gipson JD, Brindis CD, Hindin MJ, Foster DG, Dworkin SL. Development and Validation of the Sexual and Reproductive Empowerment Scale for Adolescents and Young Adults. J Adolesc Health. 2021 Jan;68(1):86-94. doi: 10.1016/j.jadohealth.2020.05.031. Epub 2020 Jul 17. PMID 32690468
- [Derived] Peitzmeier SM, Senn CY, Eliasziw M, Edwards K, Barata P, Papp LJ, Hobden KL. An Internet-Delivered Sexual Assault Resistance Intervention for Undergraduate Women (The IDEA3 Trial): Protocol for a Multisite Randomized Controlled Efficacy Trial. JMIR Res Protoc. 2025 Oct 7;14:e72087. doi: 10.2196/72087. PMID 41055953